CLINICAL TRIAL: NCT05383911
Title: Empowering Adolescents and Young Adults With Sickle Cell Disease as Partners in Treatment Decision Making (EMPOWER-AYA)
Acronym: EMPOWER-AYA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Aimee Hildenbrand, Research Scientist, Nemours Children's Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 348507
Record Dates: First submitted 2022-05-09; First posted 2022-05-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making Toolkit including VR (Experimental)
  Interventions: Behavioral: SCD Shared Decision-Making Toolkit for AYAs - including VR
- Shared Decision Making Toolkit without VR (Experimental)
  Interventions: Behavioral: SCD Shared Decision-Making Toolkit for AYAs - without VR

INTERVENTIONS:
Behavioral: SCD Shared Decision-Making Toolkit for AYAs - including VR — The SCD Shared Decision-Making Toolkit for AYAs (SDMT-AYA) targets multi-level barriers to uptake of disease-modifying therapies by providing technology-enhanced tools for: 1) clinicians (i.e., training in motivational interviewing, values elicitation, and cultural humility); 2) AYAs and caregivers (i.e., user-centered multimedia decision aids, including virtual reality, online (videos, animations, articles), and print materials); and 3) implementation (e.g., clinic audit and feedback strategies).
  Arms: Shared Decision Making Toolkit including VR
Behavioral: SCD Shared Decision-Making Toolkit for AYAs - without VR — The SCD Shared Decision-Making Toolkit for AYAs (SDMT-AYA) targets multi-level barriers to uptake of disease-modifying therapies by providing technology-enhanced tools for: 1) clinicians (i.e., training in motivational interviewing, values elicitation, and cultural humility); 2) AYAs and caregivers (i.e., user-centered multimedia decision aids, including online videos, animations, and articles as well as print materials); and 3) implementation (e.g., clinic audit and feedback strategies).
  Arms: Shared Decision Making Toolkit without VR

SUMMARY:
This study will evaluate the acceptability, feasibility, and preliminary efficacy of a shared decision making intervention for adolescents and young adults (AYAs) with sickle cell disease (SCD). 60 AYAs with SCD ages 15-25 and their caregivers and 8 SCD providers will participate in the pilot pragmatic trial. AYAs, caregivers, and providers will be recruited from Nemours Children's Hospital, Delaware (NCH-DE), Nemours Children's Hospital in Orlando, FL (NCH-ORL), and Nemours Children's Health at Wolfson Children's Hospital in Jacksonville, FL (NCH-JAX). NCH-DE participants (n=30) will receive the SDM intervention including a virtual reality patient health education component, whereas NCH-ORL and NCH-JAX participants (n=30) will receive the SDM intervention with standard patient education materials (print, video). SCD providers will be trained to use the toolkit components and will introduce decision aids during an outpatient clinic visit for AYAs who are candidates for one or more disease-modifying therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SCD ages 15-25 years receiving treatment at Nemours and their caregivers will be included. Patients must be deemed candidates for initiation of one or more disease-modifying therapies by their SCD healthcare provider.
* Nemours SCD healthcare providers will also be included.
* English language fluency is a requirement for all participants.

Exclusion Criteria:

* Patients/ caregivers who previously participated in usability testing of the intervention will be excluded.
* Patients will also be excluded if they have history of seizures, if their medical status or cognitive functioning preclude completion of interviews, or if no legal guardian is available to provide consent (for patients < 18 years).
* Providers still completing training will be excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Within 2 weeks post-intervention
  Questionnaire assessing healthcare provider perspectives on acceptability of the intervention. Total score ranges from 4-20, with higher scores indicating greater acceptability.
Patient/Caregiver Satisfaction Questionnaire | Within 2 weeks post-intervention
  Survey assessing patient/caregiver satisfaction with the intervention. Survey will be developed by the research team, and additional details will be included here once items and scoring are finalized.
Feasibility of Intervention Measure (FIM) | Within 2 weeks post-intervention
  Questionnaire assessing healthcare provider perspectives on the feasibility of the intervention. Total score ranges from 4-20, with higher scores indicating greater feasibility.
Participant Recruitment Rate | Time of enrollment through study completion, approximately 12 months
  Rate of participant enrollment and retention in the study
Shared Decision Making Questionnaire (SDM-Q-9) | Within 2 weeks post-intervention
  Questionnaire assessing patient- and caregiver-reported engagement in decision making. Total score ranges from 0 to 100, with higher scores indicating greater engagement in decision making.
Disease-Modifying Therapy Knowledge Questionnaire | Within 2 weeks post-intervention
  Questionnaire assessing patient and caregiver knowledge of disease modifying-therapies for sickle cell disease. Survey will be developed by the research team, and additional details will be included here once items and scoring are finalized.

SECONDARY OUTCOMES:
Initiation of disease-modifying therapy | Within 6 months post-intervention
  Proportion of patients who agree to initiate a disease-modifying therapy following use of the shared decision making intervention

OTHER OUTCOMES:
Acute healthcare utilization | Within 6 months post-intervention
  ED visits and hospitalizations for sickle cell-related complications during 6 months following the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Hospital, Delaware, Wilmington, Delaware, United States